CLINICAL TRIAL: NCT01328119
Title: Uremic Toxin Removal and Hemodynamics in Long-hour Hemodialysis and Hemodiafiltration; a Randomized Cross-over Study
Brief Title: Uremic Toxin Removal and Hemodynamics in Long-hour Hemodialysis and Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL34908.068.10
Record Dates: First submitted 2011-03-16; First posted 2011-04-04 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Uremic Toxins; Haemodynamic Stability

ARMS (1):
- hemodialysis patients (Other): conventional hemodialysis patients
  Interventions: Other: 4-hour HD, 4-hour HDF, 8-hour HD and 8-hour HDF

INTERVENTIONS:
Other: 4-hour HD, 4-hour HDF, 8-hour HD and 8-hour HDF — Prevalent conventional HD (CHD) patients (dialysing 3 days a week during 4 hours per dialysis session) will undergo, in random order, a mid-week 4-hour HD session, a mid-week 4-hour HDF session, a mid-week 8-hour HD session, and a mid-week 8-hour HDF session with a 2-week interval between every session to assess the influence of treatment duration and of convection on the removal of uremic toxins and on the haemodynamic responses and autonomic nervous regulation. In between the study dialysis sessions these patients will receive routine CHD treatments.

SUMMARY:
Rationale: The mortality of end-stage renal disease (ESRD) patients on dialysis remains high. This may at least be partly due to the insufficient removal of (especially protein-bound) uremic toxins which have been associated with cardiovascular morbidity and mortality. It is unknown whether the combination of long-hour haemodialysis (HD) with convection increases the removal of these toxins. Long-hour HD and long-hour haemodiafiltration (HDF) may also improve haemodynamic stability which is an important factor in treatment quality. The investigators aim to study the removal of uremic toxins in long-hour HD and HDF and to compare the haemodynamics between 4-hour and 8-hour HD and HDF.

Objectives: The primary aim is to study the removal of (especially protein-bound) uremic toxins in 4-hour and 8-hour HD and HDF. A secondary aim is to compare the haemodynamic response between 4-hour and 8-hour HD and HDF.

ELIGIBILITY:
Inclusion Criteria:

* prevalent conventional HD patients
* AV-fistula enabling double-needle vascular access with blood flow rate of at least 350 ml/min
* informed consent
* age more than 18 years

Exclusion Criteria:

* withdrawal of consent
* acute intercurrent illness (infection, malignancy, cardiovascular event, uncontrolled diabetes)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
removal of uremic toxins | before dialysis and at 15,30,60,120,240 minutes (4-hour and 8-hour sessions) and at 360 and 480 minutes (8-hour sessions)
  To measure uremic toxin and electrolyte removal, reduction ratios, dialytic clearances and mass removal in collected dialysate will be determined. Blood samples will be taken from the inlet blood lines immediately before the onset of dialysis and at 15, 30, 60, 120, 240 minutes (4-hour and 8-hour sessions) and at 360 and 480 minutes (8-hour sessions). Furthermore, ultrafiltrate and dialysate will be continuously collected in a fractionated way.

SECONDARY OUTCOMES:
haemodynamic response | every 30 minutes until end of dialysis
  BP, heart rate, heart rate variability, cardiac output and systemic vascular resistance will be measured every 30 minutes by the Task Force Monitor. Skin microcirculation will be measured with laser Doppler flowmetry every 120 min until the end of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Perl J, Chan CT. Home hemodialysis, daily hemodialysis, and nocturnal hemodialysis: Core Curriculum 2009. Am J Kidney Dis. 2009 Dec;54(6):1171-84. doi: 10.1053/j.ajkd.2009.06.038. Epub 2009 Sep 12. No abstract available. PMID 19748715